CLINICAL TRIAL: NCT00159861
Title: A Multinational, Multi-Center, Randomised, Double-Bind, Placebo-Controlled, Parallel Group Study to Assess the Safety and Efficacy of a Subject Optimised Dose of Sildenafil Citrate (20, 40, or 80 mg. Sildenafil Citrate TID) Based on the Toleration, When Used in Combination With Intravenous Prostacyclin( Epoprostenol) in the Treatment of Pulmonary Arterial Hypertension.
Brief Title: The Efficacy and Safety of Sildenafil Citrate Used in Combination With Intravenous Epoprostenol in PAH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481141; NCT00147641 (obsolete NCT alias)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2011-01-12 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Drug: Sildenafil citrate

SUMMARY:
Determination of the effects of sildenafil citrate and epoprostenol when used in combination in patients with pulmonary arterial hypertension

ELIGIBILITY:
Inclusion Criteria:

* Patients with pulmonary arterial hypertension caused by primary PAH, associated with connective tissue disease or following surgical repair of a congenital heart lesion

Exclusion Criteria:

* PH other than PAH

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2003-07; Study Completion 2006-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- United States (24):
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Torrance, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, New Orleans, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Providence, Rhode Island
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Pfizer Investigational Site, Leuven, Belgium
- Canada (4):
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Ottawa, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Montreal, Quebec
- Pfizer Investigational Site, Prague, Czechia
- Pfizer Investigational Site, Copenhagen, Denmark
- France (3):
  - Pfizer Investigational Site, Clamart
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
- Pfizer Investigational Site, Petah Tikva, Israel
- Pfizer Investigational Site, Bologna, Italy
- Netherlands (2):
  - Pfizer Investigational Site, Amsterdam
  - Pfizer Investigational Site, Nieuwegein
- Spain (2):
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
- United Kingdom (2):
  - Pfizer Investigational Site, Papworth Everard, Cambridgeshire
  - Pfizer Investigational Site, Glasgow

REFERENCES:
- [Derived] Simonneau G, Rubin LJ, Galie N, Barst RJ, Fleming TR, Frost A, Engel P, Kramer MR, Serdarevic-Pehar M, Layton GR, Sitbon O, Badesch DB; PACES Study Group. Long-term sildenafil added to intravenous epoprostenol in patients with pulmonary arterial hypertension. J Heart Lung Transplant. 2014 Jul;33(7):689-97. doi: 10.1016/j.healun.2014.02.019. Epub 2014 Feb 22. PMID 24815795
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481141&StudyName=The+Efficacy+and+Safety+of+Sildenafil+Citrate+Used+in+Combination+with+Intravenous+Epoprostenol+in+PAH+

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were entered into the open-label extension study portion upon completion of the preceding 16-week, placebo controlled core study portion or, for subjects who required a change in epoprostenol dose due to clinical deterioration, after at least 4 weeks in the core study portion.
Groups:
- Placebo: Core Study / Sildenafil: Extension Study: Core Study: Placebo (16 weeks, or at least 4 weeks for subjects who required a change in epoprostenol dose due to clinical deterioration); Extension Study: Sildenafil (until last enrolled subject completed 3 years of treatment) - initial dose 20 mg TID (3 times daily), may have been increased to 40 mg TID or 80 mg TID at discretion of Investigator
- Sildenafil: Core Study / Sildenafil: Extension Study: Core Study (16 weeks, or at least 4 weeks for subjects who required a change in epoprostenol dose due to clinical deterioration): Sildenafil 20, 40, or 80 mg TID (3 times daily) based on toleration; Extension Study (until last enrolled subject completed 3 years of treatment): Sildenafil - initial dose 20 mg TID, may have been increased to 40 mg TID or 80 mg TID at discretion of Investigator
Period: Core Study - 16 Weeks
Arm/Group | Placebo: Core Study / Sildenafil: Extension Study | Sildenafil: Core Study / Sildenafil: Extension Study
Started | 133 | 134
Treated | 131 | 134
Completed | 108 (Entered A1481153: 115; Did not enter A1481153: 16) | 122 (Entered A1481153: 127; Did not enter A1481153: 7)
Not Completed | 25 | 12
Not completed — Death | 3 | 0
Not completed — Adverse Event | 12 | 6
Not completed — Lack of Efficacy | 2 | 3
Not completed — Reason Unspecified | 5 | 3
Not completed — Subject Defaulted | 1 | 0
Not completed — Randomized but not Treated | 2 | 0
Period: Extension Study - up to 3 Years
Arm/Group | Placebo: Core Study / Sildenafil: Extension Study | Sildenafil: Core Study / Sildenafil: Extension Study
Started | 115 (Subjects may have entered extension study after 4 weeks in core study (prior to completion).) | 127 (Subjects may have entered extension study after 4 weeks in core study (prior to completion).)
Treated | 115 | 127
Completed | 53 | 56
Not Completed | 62 | 71
Not completed — Death | 24 | 28
Not completed — Adverse Event | 14 | 14
Not completed — Lack of Efficacy | 5 | 1
Not completed — Reason Unspecified | 12 | 19
Not completed — Withdrawal by Subject | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Placebo/Sildenafil: Core Study: Placebo; Extension Study: Sildenafil - initial dose 20 mg TID (3 times daily), may have been increased to 40 mg TID or 80 mg TID at discretion of Investigator
- Sildenafil/Sildenafil: Study A1481141: Sildenafil 20, 40, or 80 mg TID (3 times daily) based on toleration; Extension Study A1481153: Sildenafil - initial dose 20 mg TID, may have been increased to 40 mg TID or 80 mg TID at discretion of Investigator
- Total: Total of all reporting groups
Arm/Group | Placebo/Sildenafil | Sildenafil/Sildenafil | Total
Number analyzed (Participants) | 131 | 134 | 265
Age, Customized [Number; unit: participants]
  18 to 44 years | 47 | 54 | 101
  45 to 64 years | 73 | 64 | 137
  >= 65 years | 11 | 16 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 110 | 212
  Male | 29 | 24 | 53

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Change in Epoprostenol Dose From Baseline Maintained for 6 Months
Description: Number of subjects with changes in Epoprostenol dose from baseline maintained continuously for 6 months. Increased = Epoprostenol dose continuously more than 20% greater than core study Baseline for at least 6 months. Decrease = Epoprostenol dose continuously more than 20% less than core study Baseline for at least 6 months. No change = Epoprostenol dose change met neither Increase or Decrease criteria. Stopped = Epoprostenol dose stopped for at least 6 months.
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Month 9, and at 3-month intervals through Month 69
Population: Safety population: all subjects who took at least one dose of study medication in core study. N=number of subjects with evaluable data at core study Baseline. Includes subjects who were only treated in the core study and those who continued into the extension study.
Measure: Number; unit: participants
Groups:
- All Subjects: Core Study A1481141: Placebo or Sildenafil 20, 40, or 80 mg TID (3 times daily) based on toleration; Extension Study A1481153: Sildenafil - initial dose 20 mg TID (3 times daily), may have been increased to 40 mg TID or 80 mg TID at discretion of Investigator
Arm/Group | All Subjects
Number analyzed (Participants) | 265
participants
  Week 4: >20% Increase | 0
  Week 4: No Change | 0
  Week 4: >20% Decrease | 0
  Week 4: Stopped | 0
  Week 4: Missing | 13
  Week 8: >20% Increase | 0
  Week 8: No Change | 0
  Week 8: >20% Decrease | 0
  Week 8: Stopped | 0
  Week 8: Missing | 11
  Week 12: >20% Increase | 0
  Week 12: No Change | 0
  Week 12: >20% Decrease | 0
  Week 12: Stopped | 0
  Week 12: Missing | 14
  Week 16: >20% Increase | 0
  Week 16: No Change | 0
  Week 16: >20% Decrease | 0
  Week 16: Stopped | 0
  Week 16: Missing | 199
  Week 20: >20% Increase | 0
  Week 20: No Change | 0
  Week 20: >20% Decrease | 0
  Week 20: Stopped | 0
  Week 20: Missing | 186
  Week 24: >20% Increase | 0
  Week 24: No Change | 0
  Week 24: >20% Decrease | 0
  Week 24: Stopped | 0
  Week 24: Missing | 190
  Month 9: >20% Increase | 0
  Month 9: No Change | 0
  Month 9: >20% Decrease | 0
  Month 9: Stopped | 0
  Month 9: Missing | 174
  Month 12: >20% Increase | 4
  Month 12: No Change | 162
  Month 12: >20% Decrease | 9
  Month 12: Stopped | 0
  Month 12: Missing | 0
  Month 15: >20% Increase | 5
  Month 15: No Change | 130
  Month 15: >20% Decrease | 20
  Month 15: Stopped | 1
  Month 15: Missing | 0
  Month 18: >20% Increase | 10
  Month 18: No Change | 109
  Month 18: >20% Decrease | 27
  Month 18: Stopped | 1
  Month 18: Missing | 0
  Month 21: >20% Increase | 10
  Month 21: No Change | 105
  Month 21: >20% Decrease | 27
  Month 21: Stopped | 2
  Month 21: Missing | 0
  Month 24: >20% Increase | 15
  Month 24: No Change | 93
  Month 24: >20% Decrease | 24
  Month 24: Stopped | 2
  Month 24: Missing | 0
  Month 27: >20% Increase | 18
  Month 27: No Change | 87
  Month 27: >20% Decrease | 23
  Month 27: Stopped | 3
  Month 27: Missing | 0
  Month 30: >20% Increase | 19
  Month 30: No Change | 78
  Month 30: >20% Decrease | 23
  Month 30: Stopped | 3
  Month 30: Missing | 0
  Month 33: >20% Increase | 18
  Month 33: No Change | 76
  Month 33: >20% Decrease | 22
  Month 33: Stopped | 2
  Month 33: Missing | 0
  Month 36: >20% Increase | 20
  Month 36: No Change | 66
  Month 36: >20% Decrease | 19
  Month 36: Stopped | 4
  Month 36: Missing | 0
  Month 39: >20% Increase | 19
  Month 39: No Change | 55
  Month 39: >20% Decrease | 19
  Month 39: Stopped | 5
  Month 39: Missing | 0
  Month 42: >20% Increase | 19
  Month 42: No Change | 55
  Month 42: >20% Decrease | 18
  Month 42: Stopped | 5
  Month 42: Missing | 0
  Month 45: >20% Increase | 24
  Month 45: No Change | 51
  Month 45: >20% Decrease | 15
  Month 45: Stopped | 4
  Month 45: Missing | 0
  Month 48: >20% Increase | 23
  Month 48: No Change | 38
  Month 48: >20% Decrease | 17
  Month 48: Stopped | 5
  Month 48: Missing | 0
  Month 51: >20% Increase | 17
  Month 51: No Change | 33
  Month 51: >20% Decrease | 14
  Month 51: Stopped | 3
  Month 51: Missing | 0
  Month 54: >20% Increase | 14
  Month 54: No Change | 31
  Month 54: >20% Decrease | 14
  Month 54: Stopped | 5
  Month 54: Missing | 0
  Month 57: >20% Increase | 12
  Month 57: No Change | 27
  Month 57: >20% Decrease | 12
  Month 57: Stopped | 4
  Month 57: Missing | 0
  Month 60: >20% Increase | 12
  Month 60: No Change | 22
  Month 60: >20% Decrease | 11
  Month 60: Stopped | 2
  Month 60: Missing | 0
  Month 63: >20% Increase | 6
  Month 63: No Change | 21
  Month 63: >20% Decrease | 4
  Month 63: Stopped | 1
  Month 63: Missing | 0
  Month 66: >20% Increase | 4
  Month 66: No Change | 15
  Month 66: >20% Decrease | 2
  Month 66: Stopped | 1
  Month 66: Missing | 0
  Month 69: >20% Increase | 4
  Month 69: No Change | 9
  Month 69: >20% Decrease | 1
  Month 69: Stopped | 0
  Month 69: Missing | 0

2. Secondary Outcome: Survival Status
Description: Yearly survival status: number of subjects who survived, discontinued, and died. Analysis includes post-treatment visit data from subjects who discontinued study treatment. Time to death was taken relative to the first dose of study treatment in A1481141, and was censored on the last day the subject was known to be alive in A1481141 or A1481153.
Time Frame: 1, 2, 3, 4, and 5 years
Population: Full analysis set: all randomized and treated subjects recruited into core study. N=number of subjects with evaluable data at core study Baseline.
Measure: Number; unit: participants
Arm/Group | All Subjects
Number analyzed (Participants) | 265
participants
  1 year: Deaths | 24
  1 Year: Survived 1 Year of Study | 205
  1 Year: Discontinued before 1 Year of Study | 36
  2 Years: Deaths | 48
  2 Years: Survived 2 Years of Study | 169
  2 Years: Discontinued before 2 Years of Study | 48
  3 Years: Deaths | 64
  3 Years: Survived 3 Years of Study | 133
  3 Years: Discontinued before 3 Years of Study | 68
  4 Years: Deaths | 71
  4 Years: Survived 4 Years of Study | 88
  4 Years: Discontinued before 4 Years of Study | 75
  4 Years: Ongoing for Less than Timepoint | 26
  5 Years: Deaths | 82
  5 Years: Survived 5 Years of Study | 29
  5 Years: Discontinued before 5 Years of Study | 74
  5 Years: Ongoing for Less than Timepoint | 78
Statistical Analysis 1: Comparison: All Subjects; 1 Year: Proportion of participants who died; Test type: Superiority or Other; Kaplan-Meier estimate = 0.095, 95% CI 2-sided [0.059 to 0.132]
Statistical Analysis 2: Comparison: All Subjects; 2 Years: Proportion of participants who died; Test type: Superiority or Other; Kaplan-Meier estimate = 0.194, 95% CI 2-sided [0.144 to 0.243]
Statistical Analysis 3: Comparison: All Subjects; 3 Years: Proportion of participants who died; Test type: Superiority or Other; Kaplan-Meier estimate = 0.260, 95% CI 2-sided [0.205 to 0.315]
Statistical Analysis 4: Comparison: All Subjects; 4 Years: Proportion of participants who died; Test type: Superiority or Other; Kaplan-Meier estimate = 0.291, 95% CI 2-sided [0.234 to 0.348]
Statistical Analysis 5: Comparison: All Subjects; 5 Years: Proportion of participants who died; Test type: Superiority or Other; Kaplan-Meier estimate = 0.369, 95% CI 2-sided [0.302 to 0.437]

3. Primary Outcome: Categorized Change From Baseline in 6-Minute Walking Distance
Description: Number of subjects with categorized change in 6-minute walking distance. Distance that a subject could walk in 6-minutes at a comfortable pace with as many breaks as needed. Performed as close to trough levels of sildenafil as possible (just before dosing; at least 4 hours after the previous dose of study drug). Scores for categorized changes for missing visits were imputed as the worse score of its non-missing neighbors. If a visit was missing and there was no subsequent score, the score was coded to missing.
Time Frame: 1 Year, 2 Year, 3 Year
Population: FAS. m = meters. N=number of subjects with evaluable data at core study Baseline. Treatment groups shown by core study randomization; includes subjects who were only treated in the core study and those who continued into the extension study.
Measure: Number; unit: participants
Groups:
- Sildenafil/Sildenafil: Core Study: Sildenafil 20, 40, or 80 mg TID (3 times daily) based on toleration; Extension Study: Sildenafil - initial dose 20 mg TID, may have been increased to 40 mg TID or 80 mg TID at discretion of Investigator
Arm/Group | Placebo/Sildenafil | Sildenafil/Sildenafil
Number analyzed (Participants) | 131 | 134
participants
  1 Year: >= 60 m Improvement | 27 | 46
  1 Year: 60 - 30 m Improvement | 20 | 26
  1 Year: 30 - 0 m Improvement | 23 | 15
  1 Year: 0 - 30 m Worsening | 12 | 10
  1 Year: 30 - 60 m Worsening | 6 | 6
  1 Year: > 60 m Worsening | 6 | 6
  1 Year: Discontinued | 22 | 14
  1 Year: Died | 14 | 10
  1 Year: Missing | 1 | 1
  2 Year: >= 60 m Improvement | 23 | 44
  2 Year: 60 - 30 m Improvement | 16 | 10
  2 Year: 30 - 0 m Improvement | 15 | 8
  2 Year: 0 - 30 m Worsening | 18 | 9
  2 Year: 30 - 60 m Worsening | 2 | 7
  2 Year: > 60 m Worsening | 7 | 7
  2 Year: Discontinued | 25 | 23
  2 Year: Died | 24 | 24
  2 Year: Missing | 1 | 2
  3 Year: >= 60 m Improvement | 22 | 29
  3 Year: 60 - 30 m Improvement | 9 | 10
  3 Year: 30 - 0 m Improvement | 10 | 8
  3 Year: 0 - 30 m Worsening | 15 | 5
  3 Year: 30 - 60 m Worsening | 3 | 7
  3 Year: > 60 m Worsening | 5 | 8
  3 Year: Discontinued | 35 | 33
  3 Year: Died | 31 | 33
  3 Year: Missing | 1 | 1

4. Secondary Outcome: Change in Pulmonary Hypertension Criteria for Functional Capacity and Therapeutic Class
Description: Pulmonary hypertension (PH) criteria: Class I: PH without limitation of physical activity (PA) (no undue dyspnea, fatigue, chest pain, near syncope); Class II: PH with slight limitation in PA, comfortable at rest, ordinary PA causes undue dyspnea, fatigue, chest pain, near syncope; Class III: PH with marked limitation in PA, comfortable at rest, less than ordinary activity causes undue dyspnea, fatigue, chest pain or syncope; Class IV: PH with inability to carry out PA without symptoms, signs of right heart failure, dyspnea or fatigue may be present at rest, discomfort increased by any PA.
Time Frame: 1 Year, 2 Year, 3 Year
Population: FAS; N=number of subjects with evaluable data at core study Baseline. Treatment groups shown by core study randomization; includes subjects in core study and in extension study. Scores for categorized changes for missing visits imputed as worse score of its non-missing neighbors; missing visits with no subsequent score: score coded to missing.
Measure: Number; unit: participants
Arm/Group | Placebo/Sildenafil | Sildenafil/Sildenafil
Number analyzed (Participants) | 131 | 134
participants
  1 Year: Improved 2 Classes | 2 | 3
  1 Year: Improved 1 Class | 27 | 46
  1 Year: No Change | 59 | 57
  1 Year: Worsened 1 Class | 7 | 3
  1 Year: Worsened 2 Classes | 0 | 1
  1 Year: Discontinued | 22 | 14
  1 Year: Died | 14 | 10
  2 Year: Improved 2 Classes | 1 | 4
  2 Year: Improved 1 Class | 24 | 31
  2 Year: No Change | 50 | 47
  2 Year: Worsened 1 Class | 7 | 5
  2 Year: Worsened 2 Classes | 0 | 0
  2 Year: Discontinued | 25 | 23
  2 Year: Died | 24 | 24
  3 Year: Improved 2 Classes | 1 | 4
  3 Year: Improved 1 Class | 21 | 21
  3 Year: No Change | 39 | 37
  3 Year: Worsened 1 Class | 3 | 6
  3 Year: Worsened 2 Classes | 1 | 0
  3 Year: Discontinued | 35 | 33
  3 Year: Died | 31 | 33

5. Secondary Outcome: Change From Baseline in Medical Outcomes Study Short Form 36 (SF-36)
Description: Subject-rated measure of health status comprised of 36 items: 8 subscale scores (physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health), 2 summary scores (physical component and mental component), and a self-evaluated change in health status. Subscale and summary scores range: 0-100. Higher subscale and summary scores = better health status. Change from baseline = score at observation minus score at baseline.
Time Frame: Baseline, Month 15, Month 27, Month 39
Population: FAS. N=number of subjects with evaluable data at core study Baseline; n=number of subjects with SF-36 score at observation, Placebo, Sildenafil, respectively. Treatment groups shown by core study randomization; includes subjects who who were only treated in the core study and those who continued into the extension study. Phys = physical.
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Placebo/Sildenafil | Sildenafil/Sildenafil
Number analyzed (Participants) | 131 | 134
scores on scale
  Month 15: Physical Functioning Score (n=59, 83) | 10.5 [6.0 to 15.1] | 14.8 [10.1 to 19.4]
  Month 27: Physical Functioning Score (n=60, 62) | 9.7 [5.0 to 14.4] | 12.5 [7.1 to 17.9]
  Month 39: Physical Functioning Score (n=42, 47) | 8.9 [1.9 to 15.9] | 14.0 [7.6 to 20.4]
  Month 15: Role Limitations (phys health)(n=59, 82) | 15.7 [4.9 to 26.4] | 14.2 [3.3 to 25.2]
  Month 27: Role Limitations (phys health)(n=60, 62) | 4.6 [-8.3 to 17.5] | 2.6 [-9.8 to 14.9]
  Month 39: Role Limitations (phys health)(n=42, 47) | 4.2 [-11.0 to 19.4] | 5.1 [-9.8 to 20.1]
  Month 15: Bodily Pain Score (n=59, 82) | 10.4 [4.5 to 16.3] | 5.9 [0.3 to 11.5]
  Month 27: Bodily Pain Score (n=60, 62) | -0.1 [-6.4 to 6.3] | 4.0 [-1.8 to 9.9]
  Month 39: Bodily Pain Score (n=42, 46) | -4.9 [-13.2 to 3.4] | 3.5 [-3.4 to 10.5]
  Month 15: General Health Score (n=59, 83) | -0.2 [-5.5 to 5.2] | 10.1 [5.4 to 14.7]
  Month 27: General Health Score (n=60, 62) | 2.7 [-2.6 to 8.1] | 6.9 [2.0 to 11.7]
  Month 39: General Health Score (n=41, 47) | 3.1 [-2.6 to 8.7] | 3.4 [-2.8 to 9.7]
  Month 15: Vitality Score (n=59, 83) | 5.0 [-0.3 to 10.4] | 8.9 [3.7 to 14.0]
  Month 27: Vitality Score (n=60, 62) | 5.7 [0.8 to 10.5] | 7.2 [2.0 to 12.3]
  Month 39: Vitality Score (n=42, 47) | 6.9 [0.3 to 13.6] | 5.2 [-0.7 to 11.1]
  Month 15: Social Functioning Score (n=59, 83) | 5.9 [-2.2 to 14.1] | 5.1 [-1.2 to 11.5]
  Month 27: Social Functioning Score (n=60, 63) | 6.7 [-0.6 to 13.9] | 1.4 [-6.5 to 9.3]
  Month 39: Social Functioning Score (n=42, 47) | 2.4 [-5.9 to 10.6] | -0.8 [-9.3 to 7.7]
  Month 15: Role Limitations (Emotional) (n=59, 82) | 1.7 [-10.1 to 13.5] | 1.2 [-8.8 to 11.3]
  Month 27: Role Limitations (Emotional) (n=60, 62) | -1.7 [-13.4 to 10.0] | -7.0 [-18.1 to 4.1]
  Month 39: Role Limitations (Emotional) (n=42, 47) | 3.2 [-10.7 to 17.1] | 2.1 [-7.5 to 11.8]
  Month 15: Mental Health Score (n=59, 83) | 0.5 [-3.9 to 4.9] | 3.3 [-1.1 to 7.7]
  Month 27: Mental Health Score (n=60, 62) | 0.9 [-3.4 to 5.1] | 0.1 [-4.6 to 4.8]
  Month 39: Mental Health Score (n=42, 47) | 0.8 [-4.9 to 6.6] | 3.7 [-1.9 to 9.3]

6. Secondary Outcome: Change From Baseline in European Quality of Life Scale (EuroQol) 5-Dimensions (EQ-5D): Utility Index Score
Description: EQ-5D: subject rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state (confined to bed). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline, Month 15, Month 27, Month 39
Population: FAS. N=number of subjects with evaluable data at core study Baseline; n=number of subjects with evaluable data at observation, Placebo, Sildenafil, respectively. Treatment groups shown by core study randomization; includes subjects who who were only treated in the core study and those who continued into the extension study.
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Placebo/Sildenafil | Sildenafil/Sildenafil
Number analyzed (Participants) | 124 | 125
scores on scale
  Month 15 (n=58, 78) | 0.0505 [-0.0078 to 0.1087] | 0.0473 [-0.0065 to 0.1012]
  Month 27 (n=56, 60) | 0.0489 [-0.0146 to 0.1123] | 0.0483 [-0.0272 to 0.1237]
  Month 39 (n=40, 43) | -0.0278 [-0.1253 to 0.0697] | 0.0770 [0.0013 to 0.1526]

7. Secondary Outcome: Change From Baseline in European Quality of Life (EuroQol) Visual Analogue Scale (EQ-5D VAS): Current Health State Score
Description: EQ-5D: subject rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 (worst imaginable health state) to 100 (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline, Month 15, Month 27, Month 39
Population: FAS. N=number of subjects with evaluable data at core study Baseline; n=number of subjects with evaluable data at observation, Placebo, Sildenafil, respectively. Treatment groups shown by core study randomization; includes subjects who who were only treated in the core study and those continued into the extension study.
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Placebo/Sildenafil | Sildenafil/Sildenafil
Number analyzed (Participants) | 125 | 126
scores on scale
  Month 15 (n=57, 81) | 6.8 [2.4 to 11.1] | 12.8 [8.3 to 17.3]
  Month 27 (n=55, 60) | 5.5 [1.7 to 9.3] | 11.2 [5.9 to 16.4]
  Month 39 (n=40, 41) | 4.7 [-0.2 to 9.5] | 11.5 [5.5 to 17.5]

8. Secondary Outcome: Change From Baseline in Medical Outcomes Study Short Form 36 (SF-36): Reported Health Transition Score
Description: Subject-rated measure of health status (36 items): 8 subscale scores (physical functioning, role limitations due to physical health problems, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, mental health), 2 summary scores (physical component, mental component), and a self-evaluated change in health status. Change from Baseline in SF-36 Health Transition score at each visit. I=much better than 1 year ago; II=somewhat better than 1 year ago; III=about the same as 1 year ago; IV=somewhat worse than 1 year ago; V=much worse than 1 year ago
Time Frame: Baseline, Month 15, Month 27, Month 39
Population: FAS. N=number of subjects with evaluable data at core study Baseline. Treatment groups shown by core study randomization; includes subjects who who were only treated in the core study and those continued into the extension study. BL=Baseline.
Measure: Number; unit: participants
Arm/Group | Placebo/Sildenafil | Sildenafil/Sildenafil
Number analyzed (Participants) | 131 | 134
participants
  BL I; Month 15: I | 2 | 9
  BL I; Month 15: II | 5 | 4
  BL I; Month 15: III | 5 | 2
  BL I; Month 15: IV | 0 | 1
  BL I; Month 15: V | 0 | 0
  BL II; Month 15: I | 7 | 5
  BL II; Month 15: II | 9 | 12
  BL II; Month 15: III | 3 | 7
  BL II; Month 15: IV | 1 | 2
  BL II; Month 15: V | 0 | 0
  BL III; Month 15: I | 3 | 4
  BL III; Month 15: II | 6 | 8
  BL III; Month 15: III | 11 | 7
  BL III; Month 15: IV | 0 | 2
  BL III; Month 15: V | 0 | 0
  BL IV; Month 15: I | 2 | 5
  BL IV; Month 15: II | 0 | 3
  BL IV; Month 15: III | 2 | 3
  BL IV; Month 15: IV | 1 | 4
  BL IV; Month 15: V | 1 | 0
  BL V; Month 15: I | 0 | 1
  BL V; Month 15: II | 0 | 3
  BL V; Month 15: III | 0 | 1
  BL V; Month 15: IV | 0 | 0
  BL V; Month 15: V | 0 | 0
  Month 15: Missing Data | 73 | 51
  BL I; Month 27: I | 4 | 2
  BL I; Month 27: II | 2 | 6
  BL I; Month 27: III | 2 | 2
  BL I; Month 27: IV | 3 | 0
  BL I; Month 27: V | 0 | 0
  BL II; Month 27: I | 4 | 3
  BL II; Month 27: II | 9 | 7
  BL II; Month 27: III | 8 | 7
  BL II; Month 27: IV | 1 | 3
  BL II; Month 27: V | 0 | 0
  BL III; Month 27: I | 3 | 5
  BL III; Month 27: II | 7 | 6
  BL III; Month 27: III | 9 | 7
  BL III; Month 27: IV | 2 | 3
  BL III; Month 27: V | 0 | 0
  BL IV; Month 27: I | 1 | 1
  BL IV; Month 27: II | 1 | 3
  BL IV; Month 27: III | 1 | 3
  BL IV; Month 27: IV | 1 | 3
  BL IV; Month 27: V | 0 | 0
  BL V; Month 27: I | 0 | 1
  BL V; Month 27: II | 0 | 0
  BL V; Month 27: III | 0 | 1
  BL V; Month 27: IV | 0 | 0
  BL V; Month 27: V | 0 | 0
  Month 27: Missing Data | 73 | 71
  BL I; Month 39: I | 1 | 2
  BL I; Month 39: II | 2 | 4
  BL I; Month 39: III | 3 | 4
  BL I; Month 39: IV | 1 | 1
  BL I; Month 39: V | 0 | 0
  BL II; Month 39: I | 4 | 5
  BL II; Month 39: II | 6 | 3
  BL II; Month 39: III | 6 | 6
  BL II; Month 39: IV | 3 | 1
  BL II; Month 39: V | 0 | 0
  BL III; Month 39: I | 2 | 3
  BL III; Month 39: II | 3 | 3
  BL III; Month 39: III | 8 | 6
  BL III; Month 39: IV | 1 | 1
  BL III; Month 39: V | 0 | 0
  BL IV; Month 39: I | 0 | 0
  BL IV; Month 39: II | 1 | 0
  BL IV; Month 39: III | 0 | 2
  BL IV; Month 39: IV | 1 | 4
  BL IV; Month 39: V | 0 | 0
  BL V; Month 39: I | 0 | 1
  BL V; Month 39: II | 0 | 0
  BL V; Month 39: III | 0 | 1
  BL V; Month 39: IV | 0 | 0
  BL V; Month 39: V | 0 | 0
  Month 39: Missing Data | 89 | 87

9. Secondary Outcome: Change From Baseline in BORG Dyspnea Score
Description: BORG Dyspnea score: change from core study Baseline. Subject rating of maximum degree of dyspnea experienced at any time during the 6-Minute Walk Test. Range: 0 (no breathlessness at all) to 10 (maximum breathlessness).
Time Frame: Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24, Month 9, Month 12, Month 15, Month 18, Month 21, Month 24, Month 27, Month 30, Month 33, Month 36
Population: FAS. N=number of subjects with evaluable data at core study Baseline; n=number of subjects with evaluable data at observation, Placebo, Sildenafil, respectively. Treatment groups shown by core study randomization; includes subjects who were only treated in the core study and those who continued into the extension study.
Measure: Median (Full Range); unit: scores on scale
Groups:
- Placebo/Sildenafil: Core Study A1481141: Placebo TID (3 times daily); Extension Study A1481153: Sildenafil - initial dose 20 mg TID (3 times daily), may have been increased to 40 mg TID or 80 mg TID at discretion of Investigator
- Sldenafil/Sildenafil: Core Study A1481141: Sildenafil 20, 40, or 80 mg TID (3 times daily) based on toleration; Extension Study A1481153: Sildenafil - initial dose 20 mg TID (3 times daily), may have been increased to 40 mg TID or 80 mg TID at discretion of Investigator
Arm/Group | Placebo/Sildenafil | Sldenafil/Sildenafil
Number analyzed (Participants) | 115 | 123
scores on scale
  Week 4 (n=112, 120) | 0.0 [-9.0 to 10.0] | 0.0 [-6.0 to 4.0]
  Week 8 (n=106, 113) | 0.0 [-8.0 to 9.0] | 0.0 [-6.0 to 4.0]
  Week 12 (n=102, 108) | 0.0 [-6.0 to 4.0] | 0.0 [-7.0 to 4.0]
  Week 16 (n=95, 106) | 0.0 [-6.0 to 9.0] | 0.0 [-7.0 to 6.0]
  Week 20 (n=80, 96) | 0.0 [-8.0 to 6.0] | 0.0 [-7.0 to 4.0]
  Week 24 (n=91, 105) | 0.0 [-7.0 to 4.0] | 0.0 [-8.0 to 4.0]
  Month 9 (n=75, 98) | 0.0 [-4.0 to 4.0] | 0.0 [-8.0 to 5.0]
  Month 12 (n=72, 90) | 0.0 [-6.0 to 4.0] | 0.0 [-7.0 to 4.0]
  Month 15 (n=75, 91) | 0.0 [-6.0 to 3.0] | 0.0 [-9.0 to 4.0]
  Month 18 (n=67, 74) | 0.0 [-7.0 to 3.0] | 0.0 [-8.0 to 4.0]
  Month 21 (n=67, 79) | 0.0 [-6.0 to 3.0] | 0.0 [-7.0 to 4.0]
  Month 24 (n=68, 60) | 0.0 [-6.0 to 7.0] | 0.0 [-7.0 to 5.0]
  Month 27 (n=67, 69) | 0.0 [-4.0 to 4.0] | 0.0 [-7.0 to 3.0]
  Month 30 (n=55, 68) | 0.0 [-7.0 to 7.0] | 0.0 [-8.0 to 5.0]
  Month 33 (n=62, 65) | 0.0 [-4.0 to 7.0] | 0.0 [-7.0 to 6.0]
  Month 36 (n=51, 62) | 0.0 [-7.0 to 5.0] | 0.0 [-7.0 to 5.0]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- Placebo/Sildenafil: Core Study (16 weeks, or at least 4 weeks for subjects who required a change in epoprostenol dose due to clinical deterioration): Placebo; Extension Study (until last enrolled subject completed 3 years of treatment): Sildenafil - initial dose 20 mg TID (3 times daily), may have been increased to 40 mg TID or 80 mg TID at discretion of Investigator
- Sildenafil/Sildenafil: Core Study (16 weeks, or at least 4 weeks for subjects who required a change in epoprostenol dose due to clinical deterioration): Sildenafil 20, 40, or 80 mg TID (3 times daily) based on toleration; Extension Study (until last enrolled subject completed 3 years of treatment): Sildenafil - initial dose 20 mg TID, may have been increased to 40 mg TID or 80 mg TID at discretion of Investigator
- Placebo/Discontinued: Core Study (16 weeks, or at least 4 weeks for subjects who required a change in epoprostenol dose due to clinical deterioration): Placebo; Extension Study (until last enrolled subject completed 3 years of treatment): Discontinued
Arm/Group | Placebo/Sildenafil | Sildenafil/Sildenafil | Placebo/Discontinued
Serious Adverse Events (participants affected / at risk) | 93/115 | 104/134 | 7/16
Other Adverse Events (participants affected / at risk) | 115/115 | 134/134 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Sildenafil (N=115) | Sildenafil/Sildenafil (N=134) | Placebo/Discontinued (N=16)
Anaemia (Blood and lymphatic system disorders) | 9 | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 3 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 5 | 0
Atrial flutter (Cardiac disorders) | 1 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac arrest (Cardiac disorders) | 3 | 8 | 0
Cardiac failure (Cardiac disorders) | 6 | 5 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Cardiac valve vegetation (Cardiac disorders) | 1 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0
Electromechanical dissociation (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Palpitations (Cardiac disorders) | 2 | 2 | 0
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 16 | 13 | 2
Sinus arrest (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 5 | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 3 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 4 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 7 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 0
Ascites (Gastrointestinal disorders) | 5 | 4 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Colonic obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 0
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Femoral hernia, obstructive (Gastrointestinal disorders) | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 1 | 0
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 5 | 3 | 0
Haemorrhagic ascites (Gastrointestinal disorders) | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 2 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 6 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 3 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Proctocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 2 | 0
Retroperitoneal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 6 | 0
Asthenia (General disorders) | 1 | 1 | 0
Catheter related complication (General disorders) | 14 | 3 | 0
Catheter site erythema (General disorders) | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Catheter site inflammation (General disorders) | 0 | 1 | 0
Catheter site pain (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 9 | 3 | 0
Drug interaction (General disorders) | 1 | 2 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 0
General physical health deterioration (General disorders) | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 1
Malaise (General disorders) | 2 | 0 | 0
Oedema (General disorders) | 2 | 0 | 0
Oedema peripheral (General disorders) | 2 | 3 | 0
Pyrexia (General disorders) | 2 | 4 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 4 | 5 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Bacterial sepsis (Infections and infestations) | 0 | 0 | 1
Breast cellulitis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 5 | 2 | 0
Catheter bacteraemia (Infections and infestations) | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 15 | 17 | 0
Catheter sepsis (Infections and infestations) | 4 | 5 | 0
Catheter site cellulitis (Infections and infestations) | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 6 | 6 | 0
Cellulitis (Infections and infestations) | 1 | 4 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 0 | 0
Central line infection (Infections and infestations) | 8 | 13 | 0
Clostridial infection (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 4 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1 | 0
Endocarditis staphylococcal (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 2 | 0
Implant site infection (Infections and infestations) | 0 | 1 | 0
Infusion site infection (Infections and infestations) | 1 | 0 | 0
Listeriosis (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Oropharyngeal candidiasis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 11 | 12 | 0
Sepsis (Infections and infestations) | 9 | 6 | 0
Septic shock (Infections and infestations) | 0 | 2 | 0
Serratia infection (Infections and infestations) | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1 | 0
Complications of transplant surgery (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Device breakage (Injury, poisoning and procedural complications) | 3 | 0 | 0
Device failure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Device malfunction (Injury, poisoning and procedural complications) | 0 | 3 | 0
Device migration (Injury, poisoning and procedural complications) | 5 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bleeding time prolonged (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0
Body temperature increased (Investigations) | 1 | 0 | 0
Electrocardiogram change (Investigations) | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0
Pulmonary arterial pressure increased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 2 | 0
Diplegia (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Facial palsy (Nervous system disorders) | 0 | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 3 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 8 | 4 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Transverse sinus thrombosis (Nervous system disorders) | 0 | 1 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 2 | 0
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 2 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine enlargement (Reproductive system and breast disorders) | 1 | 0 | 0
Alveolitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 14 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 7 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 15 | 22 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cardiac ablation (Surgical and medical procedures) | 1 | 0 | 0
Catheter placement (Surgical and medical procedures) | 1 | 1 | 0
Drug therapy changed (Surgical and medical procedures) | 0 | 1 | 0
Haematoma evacuation (Surgical and medical procedures) | 1 | 0 | 0
Indwelling catheter management (Surgical and medical procedures) | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 2 | 0
Hypotension (Vascular disorders) | 5 | 4 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0
Shock (Vascular disorders) | 3 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Vasodilatation (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo/Sildenafil (N=115) | Sildenafil/Sildenafil (N=134) | Placebo/Discontinued (N=16)
Anaemia (Blood and lymphatic system disorders) | 23 | 17 | 0
Coagulopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 | 7 | 0
Leukocytosis (Blood and lymphatic system disorders) | 3 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 7 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 5 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 4 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 3 | 2 | 0
Paratracheal lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Splenic granuloma (Blood and lymphatic system disorders) | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 3 | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 17 | 10 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 2 | 0 | 0
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 3 | 0
Bradycardia (Cardiac disorders) | 3 | 2 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Cardiac failure high output (Cardiac disorders) | 0 | 1 | 0
Cardiac flutter (Cardiac disorders) | 0 | 2 | 1
Cardiac valve vegetation (Cardiac disorders) | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 1
Cardiomegaly (Cardiac disorders) | 1 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 2 | 0
Cyanosis (Cardiac disorders) | 2 | 4 | 0
Extrasystoles (Cardiac disorders) | 1 | 3 | 0
Hepatojugular reflux (Cardiac disorders) | 3 | 1 | 0
Palpitations (Cardiac disorders) | 33 | 32 | 0
Pericardial cyst (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 3 | 7 | 0
Pulmonary valve disease (Cardiac disorders) | 0 | 1 | 0
Pulmonary valve incompetence (Cardiac disorders) | 1 | 0 | 0
Right ventricular failure (Cardiac disorders) | 6 | 3 | 0
Right ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 3 | 0
Supraventricular tachycardia (Cardiac disorders) | 4 | 3 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 9 | 10 | 0
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 0
Colour blindness (Congenital, familial and genetic disorders) | 0 | 1 | 0
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 2 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 2 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 0 | 1 | 0
Ear disorder (Ear and labyrinth disorders) | 2 | 0 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 4 | 2 | 0
Ear pruritus (Ear and labyrinth disorders) | 1 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 2 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 3 | 0
Vertigo (Ear and labyrinth disorders) | 9 | 9 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 3 | 0
Adrenal cyst (Endocrine disorders) | 1 | 0 | 0
Adrenal mass (Endocrine disorders) | 2 | 0 | 0
Autoimmune thyroiditis (Endocrine disorders) | 1 | 0 | 0
Basedow's disease (Endocrine disorders) | 1 | 1 | 0
Goitre (Endocrine disorders) | 1 | 6 | 0
Growth hormone deficiency (Endocrine disorders) | 1 | 0 | 0
Hyperadrenalism (Endocrine disorders) | 0 | 1 | 0
Hyperprolactinaemia (Endocrine disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 3 | 5 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0 | 0
Hypothalamo-pituitary disorder (Endocrine disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 4 | 3 | 0
Thyroid disorder (Endocrine disorders) | 1 | 1 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0
Toxic nodular goitre (Endocrine disorders) | 0 | 1 | 0
Abnormal sensation in eye (Eye disorders) | 1 | 1 | 0
Blepharitis (Eye disorders) | 1 | 2 | 0
Cataract (Eye disorders) | 3 | 2 | 0
Chalazion (Eye disorders) | 1 | 0 | 0
Choroidal detachment (Eye disorders) | 0 | 1 | 0
Chromatopsia (Eye disorders) | 1 | 4 | 0
Conjunctival haemorrhage (Eye disorders) | 4 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 2 | 3 | 0
Conjunctivitis (Eye disorders) | 1 | 3 | 0
Cyanopsia (Eye disorders) | 2 | 4 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 2 | 1 | 0
Dry eye (Eye disorders) | 1 | 4 | 0
Eye disorder (Eye disorders) | 0 | 1 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0
Eye inflammation (Eye disorders) | 0 | 2 | 0
Eye irritation (Eye disorders) | 2 | 1 | 0
Eye oedema (Eye disorders) | 0 | 1 | 0
Eye pain (Eye disorders) | 2 | 3 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 1 | 2 | 0
Eyelid oedema (Eye disorders) | 2 | 2 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 3 | 1 | 0
Myodesopsia (Eye disorders) | 0 | 1 | 0
Myopia (Eye disorders) | 1 | 0 | 0
Night blindness (Eye disorders) | 1 | 1 | 0
Ocular hyperaemia (Eye disorders) | 2 | 5 | 0
Ocular icterus (Eye disorders) | 0 | 1 | 0
Photophobia (Eye disorders) | 6 | 4 | 0
Photopsia (Eye disorders) | 1 | 3 | 0
Presbyopia (Eye disorders) | 0 | 1 | 0
Retinal degeneration (Eye disorders) | 0 | 1 | 0
Retinal disorder (Eye disorders) | 0 | 2 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0
Scleritis (Eye disorders) | 0 | 1 | 0
Venous stasis retinopathy (Eye disorders) | 0 | 1 | 0
Vision blurred (Eye disorders) | 9 | 11 | 0
Visual acuity reduced (Eye disorders) | 2 | 0 | 0
Visual brightness (Eye disorders) | 0 | 1 | 0
Visual impairment (Eye disorders) | 3 | 6 | 0
Xanthopsia (Eye disorders) | 1 | 2 | 0
Xerophthalmia (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 7 | 5 | 0
Abdominal distension (Gastrointestinal disorders) | 15 | 13 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 13 | 22 | 3
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 17 | 13 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1
Anal inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Anal pruritus (Gastrointestinal disorders) | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 18 | 12 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 0 | 2 | 0
Breath odour (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 7 | 11 | 1
Dental caries (Gastrointestinal disorders) | 3 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 54 | 64 | 5
Diverticulum (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 9 | 11 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 20 | 32 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 0 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 3 | 3 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 6 | 5 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 3 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal telangiectasia (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 | 13 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 2 | 3 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 3 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0 | 0
Intestinal functional disorder (Gastrointestinal disorders) | 1 | 0 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 2 | 0 | 0
Leukoplakia oral (Gastrointestinal disorders) | 1 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 48 | 63 | 4
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal dilatation (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal disorder (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal hypomotility (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 5 | 2 | 0
Oral disorder (Gastrointestinal disorders) | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic calcification (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic disorder (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 1 | 0
Polyp colorectal (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 3 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0
Reflux oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 1 | 0
Salivary duct obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0
Tongue discolouration (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 2 | 3 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 31 | 41 | 2
Vomiting projectile (Gastrointestinal disorders) | 0 | 1 | 0
Abasia (General disorders) | 1 | 0 | 0
Asthenia (General disorders) | 13 | 21 | 1
Catheter related complication (General disorders) | 11 | 10 | 0
Catheter site discharge (General disorders) | 6 | 6 | 0
Catheter site erosion (General disorders) | 0 | 1 | 0
Catheter site erythema (General disorders) | 3 | 6 | 0
Catheter site haematoma (General disorders) | 1 | 1 | 0
Catheter site haemorrhage (General disorders) | 4 | 7 | 0
Catheter site inflammation (General disorders) | 4 | 1 | 0
Catheter site oedema (General disorders) | 2 | 0 | 0
Catheter site pain (General disorders) | 3 | 4 | 0
Catheter site rash (General disorders) | 0 | 3 | 0
Catheter site related reaction (General disorders) | 2 | 4 | 0
Catheter thrombosis (General disorders) | 0 | 1 | 0
Chest discomfort (General disorders) | 10 | 13 | 1
Chest pain (General disorders) | 26 | 36 | 0
Chills (General disorders) | 7 | 11 | 0
Discomfort (General disorders) | 0 | 2 | 0
Early satiety (General disorders) | 1 | 0 | 0
Energy increased (General disorders) | 1 | 0 | 0
Exercise tolerance decreased (General disorders) | 0 | 1 | 0
Face oedema (General disorders) | 1 | 2 | 0
Fatigue (General disorders) | 44 | 56 | 4
Feeling cold (General disorders) | 5 | 2 | 0
Feeling hot (General disorders) | 1 | 1 | 0
Feeling jittery (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 2 | 1 | 0
Hyperthermia (General disorders) | 1 | 1 | 0
Hypothermia (General disorders) | 0 | 1 | 0
Ill-defined disorder (General disorders) | 3 | 1 | 0
Implant site discharge (General disorders) | 1 | 0 | 0
Implant site reaction (General disorders) | 0 | 1 | 0
Implant site ulcer (General disorders) | 1 | 0 | 0
Inflammation (General disorders) | 0 | 1 | 0
Influenza like illness (General disorders) | 7 | 2 | 0
Infusion site induration (General disorders) | 1 | 0 | 0
Infusion site pain (General disorders) | 1 | 1 | 0
Infusion site reaction (General disorders) | 1 | 1 | 0
Infusion site vesicles (General disorders) | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 2 | 0
Irritability (General disorders) | 2 | 2 | 0
Malaise (General disorders) | 5 | 8 | 0
Mass (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 16 | 25 | 1
Oedema peripheral (General disorders) | 37 | 38 | 1
Pain (General disorders) | 11 | 12 | 1
Pitting oedema (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 23 | 16 | 0
Sensation of blood flow (General disorders) | 0 | 1 | 0
Sensation of foreign body (General disorders) | 0 | 1 | 0
Temperature intolerance (General disorders) | 1 | 1 | 0
Tenderness (General disorders) | 2 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0
Unevaluable event (General disorders) | 0 | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 1 | 1
Hepatic congestion (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 0 | 2 | 0
Hepatic lesion (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 5 | 13 | 2
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Portal hypertension (Hepatobiliary disorders) | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 3 | 0
Multiple allergies (Immune system disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 3 | 2 | 0
Abscess (Infections and infestations) | 1 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 2 | 0
Bacterial infection (Infections and infestations) | 1 | 2 | 0
Body tinea (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 15 | 24 | 0
Bronchopneumonia (Infections and infestations) | 0 | 2 | 0
Candidiasis (Infections and infestations) | 0 | 1 | 1
Catheter related infection (Infections and infestations) | 18 | 18 | 0
Catheter sepsis (Infections and infestations) | 4 | 1 | 0
Catheter site cellulitis (Infections and infestations) | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 14 | 6 | 0
Cellulitis (Infections and infestations) | 6 | 6 | 0
Central line infection (Infections and infestations) | 9 | 9 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 1 | 0
Conjunctivitis infective (Infections and infestations) | 0 | 1 | 0
Conjunctivitis viral (Infections and infestations) | 1 | 1 | 0
Cystitis (Infections and infestations) | 2 | 2 | 0
Dacryocanaliculitis (Infections and infestations) | 0 | 1 | 0
Device related infection (Infections and infestations) | 3 | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 2 | 1
Ear lobe infection (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 2 | 0 | 0
Eye infection (Infections and infestations) | 2 | 2 | 0
Eye infection bacterial (Infections and infestations) | 0 | 1 | 0
Fungal infection (Infections and infestations) | 2 | 1 | 0
Furuncle (Infections and infestations) | 2 | 0 | 0
Gastroenteritis (Infections and infestations) | 5 | 8 | 0
Gastroenteritis viral (Infections and infestations) | 6 | 3 | 0
Genital herpes (Infections and infestations) | 1 | 0 | 0
Helicobacter infection (Infections and infestations) | 1 | 0 | 0
Hepatitis A (Infections and infestations) | 0 | 1 | 0
Herpes simplex (Infections and infestations) | 2 | 1 | 0
Herpes zoster (Infections and infestations) | 6 | 4 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0
Infected sebaceous cyst (Infections and infestations) | 0 | 1 | 0
Infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 13 | 15 | 0
Injection site infection (Infections and infestations) | 0 | 1 | 0
Localised infection (Infections and infestations) | 5 | 3 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 2 | 0
Lung infection (Infections and infestations) | 2 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 1 | 0
Moraxella infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 21 | 18 | 1
Onychomycosis (Infections and infestations) | 1 | 3 | 0
Oral candidiasis (Infections and infestations) | 6 | 2 | 0
Oral fungal infection (Infections and infestations) | 2 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0
Otitis externa (Infections and infestations) | 1 | 1 | 0
Otitis media (Infections and infestations) | 2 | 6 | 0
Parotitis (Infections and infestations) | 1 | 0 | 0
Periorbital infection (Infections and infestations) | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 1 | 2 | 0
Pharyngitis bacterial (Infections and infestations) | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 2 | 4 | 0
Pneumonia (Infections and infestations) | 6 | 3 | 1
Pulmonary mycosis (Infections and infestations) | 0 | 1 | 0
Rash pustular (Infections and infestations) | 2 | 0 | 0
Respiratory tract infection (Infections and infestations) | 5 | 4 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1
Septic embolus (Infections and infestations) | 0 | 1 | 1
Sinusitis (Infections and infestations) | 16 | 17 | 0
Skin infection (Infections and infestations) | 2 | 2 | 0
Sputum purulent (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 2 | 0
Tooth abscess (Infections and infestations) | 1 | 2 | 0
Tooth infection (Infections and infestations) | 0 | 3 | 0
Tracheitis (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 39 | 54 | 1
Urethritis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 12 | 11 | 0
Viral infection (Infections and infestations) | 3 | 3 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 3 | 3 | 0
Accidental exposure (Injury, poisoning and procedural complications) | 1 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 2 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Chillblains (Injury, poisoning and procedural complications) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 8 | 14 | 0
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Device breakage (Injury, poisoning and procedural complications) | 1 | 7 | 0
Device failure (Injury, poisoning and procedural complications) | 1 | 1 | 0
Device malfunction (Injury, poisoning and procedural complications) | 0 | 2 | 0
Device migration (Injury, poisoning and procedural complications) | 1 | 1 | 0
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 2 | 3 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 2 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incorrect dose administered (Injury, poisoning and procedural complications) | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 4 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 4 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Medical device complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Mouth injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 2 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Periorbital haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 3 | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 2 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Antinuclear antibody positive (Investigations) | 0 | 2 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Biopsy lymph gland (Investigations) | 1 | 0 | 0
Blood albumin decreased (Investigations) | 1 | 0 | 0
Blood albumin increased (Investigations) | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 0
Blood bicarbonate decreased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 1 | 0
Blood calcium decreased (Investigations) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 5 | 3 | 0
Blood culture positive (Investigations) | 1 | 1 | 0
Blood folate decreased (Investigations) | 0 | 1 | 0
Blood glucose decreased (Investigations) | 1 | 2 | 0
Blood glucose increased (Investigations) | 3 | 1 | 0
Blood iron decreased (Investigations) | 2 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 1 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0
Blood potassium decreased (Investigations) | 3 | 5 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Blood pressure decreased (Investigations) | 1 | 0 | 0
Blood pressure diastolic decreased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0
Blood pressure systolic decreased (Investigations) | 0 | 1 | 0
Blood prolactin decreased (Investigations) | 1 | 0 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 0
Blood sodium increased (Investigations) | 2 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 1 | 0
Blood urea increased (Investigations) | 3 | 5 | 0
Blood uric acid increased (Investigations) | 1 | 1 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Body temperature increased (Investigations) | 2 | 2 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0
Carbon dioxide decreased (Investigations) | 0 | 1 | 0
Cardiac index decreased (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 6 | 3 | 0
Cardiac output increased (Investigations) | 0 | 1 | 0
Cardioactive drug level below therapeutic (Investigations) | 1 | 0 | 0
Cardioactive drug level decreased (Investigations) | 1 | 0 | 0
Cardioactive drug level increased (Investigations) | 1 | 1 | 0
Catheterisation cardiac abnormal (Investigations) | 0 | 1 | 0
Chest X-ray abnormal (Investigations) | 0 | 1 | 0
Coagulation test abnormal (Investigations) | 0 | 1 | 0
Coagulation time prolonged (Investigations) | 1 | 1 | 0
Computerised tomogram abdomen abnormal (Investigations) | 1 | 0 | 0
Computerised tomogram thorax abnormal (Investigations) | 0 | 1 | 0
Drug level increased (Investigations) | 1 | 0 | 0
Electrocardiogram change (Investigations) | 1 | 0 | 0
Exercise test abnormal (Investigations) | 1 | 1 | 0
Gallop rhythm present (Investigations) | 1 | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0
Haematocrit increased (Investigations) | 2 | 1 | 0
Haemoglobin decreased (Investigations) | 4 | 1 | 0
Haemoglobin increased (Investigations) | 2 | 1 | 0
Heart rate decreased (Investigations) | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 4 | 0
Heart rate irregular (Investigations) | 0 | 1 | 0
Heart sounds abnormal (Investigations) | 3 | 1 | 0
Helicobacter pylori identification test positive (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 0 | 0
International normalised ratio decreased (Investigations) | 1 | 2 | 0
International normalised ratio increased (Investigations) | 8 | 13 | 0
Intraocular pressure increased (Investigations) | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 2 | 3 | 0
Liver scan abnormal (Investigations) | 1 | 0 | 0
Low density lipoprotein increased (Investigations) | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 2 | 0
Mean cell haemoglobin decreased (Investigations) | 0 | 1 | 0
Mean cell volume decreased (Investigations) | 1 | 1 | 0
Medical observation (Investigations) | 0 | 1 | 0
Neutrophil count increased (Investigations) | 0 | 2 | 0
Occult blood (Investigations) | 0 | 1 | 0
Occult blood positive (Investigations) | 0 | 2 | 0
Oxygen consumption increased (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 2 | 4 | 0
Platelet count decreased (Investigations) | 6 | 2 | 0
Platelet function test abnormal (Investigations) | 1 | 0 | 0
Protein total decreased (Investigations) | 1 | 0 | 0
Protein total increased (Investigations) | 0 | 2 | 0
Protein urine (Investigations) | 0 | 1 | 0
Protein urine present (Investigations) | 0 | 1 | 0
Pulmonary arterial pressure increased (Investigations) | 1 | 0 | 0
Pulmonary arterial wedge pressure increased (Investigations) | 0 | 1 | 0
Pulmonary function challenge test abnormal (Investigations) | 0 | 1 | 0
Pulse pressure decreased (Investigations) | 0 | 1 | 0
Red blood cell count increased (Investigations) | 0 | 1 | 0
Red cell distribution width increased (Investigations) | 0 | 1 | 0
Smear cervix abnormal (Investigations) | 0 | 1 | 0
Spleen scan abnormal (Investigations) | 1 | 0 | 0
Sputum culture positive (Investigations) | 0 | 1 | 0
Thyroid function test abnormal (Investigations) | 1 | 1 | 0
Thyroxine (Investigations) | 1 | 0 | 0
Thyroxine increased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Urine output decreased (Investigations) | 1 | 3 | 0
Venous pressure jugular increased (Investigations) | 5 | 3 | 0
Weight decreased (Investigations) | 15 | 15 | 0
Weight increased (Investigations) | 15 | 11 | 1
White blood cell count decreased (Investigations) | 0 | 2 | 0
White blood cell count increased (Investigations) | 1 | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 10 | 18 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 8 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 4 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 3 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 4 | 0
Gout (Metabolism and nutrition disorders) | 7 | 3 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 3 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 18 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 2 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 | 2 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 25 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 25 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Bone swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursa disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 6 | 3 | 0
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Mastication disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 11 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 8 | 6 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 15 | 13 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 16 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3 | 6 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 43 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 20 | 22 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast cancer female (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Juvenile melanoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Myolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Amnesia (Nervous system disorders) | 1 | 3 | 0
Aphonia (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Burning sensation (Nervous system disorders) | 2 | 2 | 0
Carpal tunnel syndrome (Nervous system disorders) | 2 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Coma (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0
Dementia (Nervous system disorders) | 1 | 0 | 0
Diabetic hyperosmolar coma (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 39 | 59 | 5
Dizziness exertional (Nervous system disorders) | 1 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 1 | 0
Dysgeusia (Nervous system disorders) | 5 | 4 | 0
Dysphasia (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Formication (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 75 | 91 | 3
Hemianopia (Nervous system disorders) | 0 | 1 | 0
Hyperaesthesia (Nervous system disorders) | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 8 | 8 | 0
Hypogeusia (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 3 | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 4 | 5 | 0
Migraine with aura (Nervous system disorders) | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Neuritis (Nervous system disorders) | 0 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 0
Paraesthesia (Nervous system disorders) | 5 | 6 | 0
Poor quality sleep (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 5 | 6 | 0
Restless legs syndrome (Nervous system disorders) | 4 | 1 | 0
Sciatica (Nervous system disorders) | 3 | 2 | 0
Sinus headache (Nervous system disorders) | 2 | 2 | 0
Somnolence (Nervous system disorders) | 1 | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0 | 0
Spinal cord disorder (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 9 | 10 | 1
Tension headache (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 2 | 0
Transverse sinus thrombosis (Nervous system disorders) | 0 | 1 | 0
Tremor (Nervous system disorders) | 3 | 5 | 0
Affect lability (Psychiatric disorders) | 0 | 2 | 0
Anger (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 13 | 18 | 0
Confusional state (Psychiatric disorders) | 4 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 1 | 0
Depression (Psychiatric disorders) | 19 | 18 | 1
Disturbance in sexual arousal (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 15 | 17 | 0
Mental status changes (Psychiatric disorders) | 2 | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0
Nervousness (Psychiatric disorders) | 3 | 1 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 2 | 0 | 0
Paranoia (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0
Albuminuria (Renal and urinary disorders) | 0 | 1 | 0
Azotaemia (Renal and urinary disorders) | 1 | 2 | 0
Dysuria (Renal and urinary disorders) | 3 | 4 | 0
Haematuria (Renal and urinary disorders) | 3 | 4 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 2 | 0
Nocturia (Renal and urinary disorders) | 5 | 6 | 0
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0
Renal cyst (Renal and urinary disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 7 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 2 | 0
Stress urinary incontinence (Renal and urinary disorders) | 1 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1 | 1 | 0
Breast calcifications (Reproductive system and breast disorders) | 1 | 0 | 0
Breast disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Breast enlargement (Reproductive system and breast disorders) | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 2 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 2 | 1 | 0
Breast swelling (Reproductive system and breast disorders) | 0 | 1 | 0
Breast tenderness (Reproductive system and breast disorders) | 0 | 2 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Cervix disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 2 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 2 | 0
Endometrial disorder (Reproductive system and breast disorders) | 0 | 1 | 0
Endometrial hypertrophy (Reproductive system and breast disorders) | 0 | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Erection increased (Reproductive system and breast disorders) | 1 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 2 | 1 | 0
Male sexual dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0
Menopausal symptoms (Reproductive system and breast disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 2 | 2 | 0
Menstruation delayed (Reproductive system and breast disorders) | 0 | 1 | 0
Menstruation irregular (Reproductive system and breast disorders) | 1 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 2 | 3 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0
Spontaneous penile erection (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular mass (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine inflammation (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine mass (Reproductive system and breast disorders) | 1 | 0 | 0
Uterine pain (Reproductive system and breast disorders) | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 3 | 3 | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 40 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 62 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 8 | 12 | 0
Dyspnoea paroxysmal nocturnal (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 21 | 36 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 11 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 18 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 9 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary artery aneurysm (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 15 | 11 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary vascular resistance abnormality (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 6 | 7 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Reproductive system and breast disorders) | 0 | 2 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 9 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 3 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 7 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Blood blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 4 | 7 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 | 10 | 0
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 7 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 11 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 32 | 31 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 4 | 3 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 3 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 5 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Skin nodule (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 | 2 | 0
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Subcutaneous nodule (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Telangiectasia (Skin and subcutaneous tissue disorders) | 8 | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 5 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Artificial crown procedure (Surgical and medical procedures) | 1 | 0 | 0
Cervical polypectomy (Surgical and medical procedures) | 0 | 1 | 0
Eye operation (Surgical and medical procedures) | 0 | 1 | 0
Haematoma evacuation (Surgical and medical procedures) | 1 | 0 | 0
Incisional hernia repair (Surgical and medical procedures) | 1 | 0 | 0
Intravenous catheter management (Surgical and medical procedures) | 0 | 1 | 0
Uterine polypectomy (Surgical and medical procedures) | 1 | 0 | 0
Angiopathy (Vascular disorders) | 1 | 1 | 0
Arterial disorder (Vascular disorders) | 1 | 0 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 35 | 45 | 2
Haematoma (Vascular disorders) | 6 | 4 | 0
Haemorrhage (Vascular disorders) | 4 | 1 | 0
Hot flush (Vascular disorders) | 9 | 6 | 1
Hypertension (Vascular disorders) | 2 | 3 | 0
Hypotension (Vascular disorders) | 17 | 18 | 0
Intermittent claudication (Vascular disorders) | 0 | 2 | 0
Jugular vein distension (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 1 | 0
Pallor (Vascular disorders) | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 1
Phlebitis (Vascular disorders) | 2 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 2 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 1 | 4 | 0
Vasculitis (Vascular disorders) | 0 | 1 | 0
Vasodilatation (Vascular disorders) | 2 | 3 | 0
Venous insufficiency (Vascular disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other